CLINICAL TRIAL: NCT01139671
Title: Comparison of Sufentanil and Remifentanil Infusion During General Anaesthesia for Removal of Wisdom Teeth in Ambulatory Surgery
Acronym: SUF-REM-DDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0074; 2010-018751-10 (EudraCT Number)
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Tooth Extractions
Keywords: Remifentanil; Sufentanil; Surgical removal of three to four wisdom teeth; General anaesthesia; Ambulatory oral surgery; Target Controlled Infusion (TCI); Opioid induced hyperalgesia; Postoperative nausea and vomiting; Postoperative Morphine consumption; Under General anaesthesia; In Ambulatory surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Remifentanil — Wisdom teeth removal under general anaesthesia is usually suitable for ambulatory surgery.
  The choice of opioid in dental day surgery is based on the need for a rapid and full recovery, as well as less morphine administration. Whether remifentanil can achieve these goals remains to be proved, especially regarding remifentanil-induced hyperalgesia, the potential prolonged Post Anesthesia Care Unit (PACU) stay, or remifentanil-induced workload for nurses.

SUMMARY:
Wisdom teeth removal under general anaesthesia is usually suitable for ambulatory surgery.

The choice of opioid in dental day surgery is based on the need for a rapid and full recovery, as well as less morphine administration. Whether remifentanil can achieve these goals remains to be proved, especially regarding remifentanil-induced hyperalgesia, the potential prolonged Post Anesthesia Care Unit (PACU) stay, or remifentanil-induced workload for nurses.

DETAILED DESCRIPTION:
Patients will be enrolled during the preoperative anaesthetic assessment. Premedication will be achieved with oral administration of hydroxyzine 1 mg/kg the morning before surgery.

The induction of general anaesthesia will be achieved using TARGET CONTROLLED INFUSION (TCI) of propofol associated to TCI of remifentanil or sufentanil, depending on randomization.

The conditions of endotracheal intubation will be evaluated by the Percentage Of Glottic Opening Score (POGO) and the Cormack and Lehane Score.

Mechanical volume-controled ventilation will aim to maintain normocapnia. The baseline inspiratory gas will be a mixture of 45% oxygen and 55% nitrous oxide.

Bispectral Index recording and vital signs monitoring (heart rate and arterial blood pressure) will be used to monitor the depth of anaesthesia.

Dexamethasone 0.3 mg/kg will be administered after induction of general anaesthesia as part of our routine practice.

Patients will be extubated as soon as possible after the end of the surgery and transferred to the PACU.

Nurses in charge patients included in the study will be blinded to the opiod agent administered peroperatively.

Postoperative pain will be assessed using the simple numeric scale. A pain score above 3/10 will prompt the intravenous administration of titrated morphine chlorhydrate, as guided by a written protocol.

Patient will be transferred from the PACU to the ambulatory surgery unit when the Aldrete score is greater or equal to 9. Every patient included will received 1 gr of intravenous paracetamol two hours after the arrival hour in the PACU.

Pain monitoring will be continued in the ambulatory surgery unit, and morphine chlorhydrate will be orally administered (10 mg) if pain score is above 3/10.

Post anaesthetic discharge for home readiness will be given when the Post Anesthetic Discharge Scoring System (PADSS) is greater or equal to 9.

48 hours after the surgery, one of us, blinded to the opiod agent received by the patient, will contact every included patient by phone, in order to evaluate postoperative pain, potential side effects including nausea and vomiting, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* -age between 15 and 35 years old
* American Society of Anaesthesiologists (ASA) physical status I or II
* Surgical removal of three to four wisdom teeth
* general anaesthesia
* Ambulatory surgery

Exclusion Criteria:

* Obesity (Body mass index > 30 kg.m-²)
* Pregnancy
* Contraindication for nitrous oxide inhalation
* Patient refusal

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in Post Anaesthesia Care Unit ( with intravenous titration given by nurse) | 48 h after the surgery

SECONDARY OUTCOMES:
- Postoperative pain (measured by the numeric pain intensity scale) | 48 h after the surgery
patient's satisfaction | 48 h after the surgery
Length of stay in Post Anaesthesia Care Unit and in ambulatory surgery unit | 48 h after the surgery
- Occurrence of postoperative nausea and vomiting | 48 h after the surgery
additional workload for nurses | 48 h after the surgery
postoperative analgesic requirement in the first 48 hours after surgery | 48 h after the surgery
percentage of Glottic opening (POGO) score, Cormack-Lehane grading | 48 h after the surgery
tolerance of the procedure | 48 h after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Gonnu-Levallois, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France